CLINICAL TRIAL: NCT07289633
Title: Evaluation of the Effect of Resin-Based and Bioceramic Sealers on Postoperative Pain in Mandibular Molars With Asymptomatic Apical Periodontitis Treated in a Single Visit
Brief Title: Evaluation of Postoperative Pain After Using Resin-Based and Bioceramic Sealers in Mandibular Molars With Asymptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZİZ ŞAHİN ERDOĞAN (Other)
Responsible Party: Sponsor-Investigator, AZİZ ŞAHİN ERDOĞAN, Assistant Professor of Endodontics, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2ATA.0.01.00/559
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Asymptomatic Apical Periodontitis
Keywords: Root Canal Treatment; Postoperative Pain; BioRoot RCS; AH Plus; Mandibular Molars
MeSH Terms: conditions — Pain, Postoperative | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are randomly allocated to one of two treatment groups receiving either a bioceramic-based sealer (BioRoot RCS) or a resin-based sealer (AH Plus) during single-visit root canal treatment.
Who Masked: Participant
Masking Description: his study uses a single-blind masking design. Participants are blinded to the type of root canal sealer used during treatment, but the care provider performing the procedure is not blinded. Postoperative pain is self-reported by participants using a standardized pain scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioRoot RCS Group (Experimental): Single-visit root canal treatment using BioRoot RCS (bioceramic sealer)
  Interventions: Other: BioRoot RCS
- AH Plus Group (Active Comparator): Single-visit root canal treatment using AH Plus (resin-based sealer)
  Interventions: Other: AH Plus

INTERVENTIONS:
Other: BioRoot RCS — Single-visit root canal treatment was performed on mandibular molar teeth diagnosed with asymptomatic apical periodontitis. After shaping and irrigation, the canals were obturated using the BioRoot RCS bioceramic-based sealer with a single-cone technique. No additional medicament or adjunctive procedure was used.
  Arms: BioRoot RCS Group
Other: AH Plus — Single-visit root canal treatment was performed on mandibular molar teeth diagnosed with asymptomatic apical periodontitis. After shaping and irrigation, the canals were obturated using the AH Plus resin-based sealer with a single-cone technique. No additional medicament or adjunctive procedure was used.
  Arms: AH Plus Group

SUMMARY:
This study aims to evaluate the effect of two different root canal sealers-BioRoot RCS (a bioceramic-based sealer) and AH Plus (a resin-based sealer)-on postoperative pain following single-visit root canal treatment in mandibular first and second molars diagnosed with asymptomatic apical periodontitis. Postoperative pain levels will be assessed at multiple time intervals to determine whether the type of canal sealer influences patient discomfort after treatment.

DETAILED DESCRIPTION:
Asymptomatic apical periodontitis is a common condition requiring root canal treatment, and postoperative pain is an important outcome that affects patient comfort and clinical decision-making. Root canal sealers play a critical role in the success of endodontic therapy, and their physical and biological properties may influence postoperative symptoms.

This study compares a bioceramic-based sealer (BioRoot RCS) and a resin-based sealer (AH Plus) in patients receiving single-visit root canal treatment for mandibular first and second molars with asymptomatic apical periodontitis. Participants will be randomly assigned to one of the two sealer groups. Pain intensity will be recorded using a validated pain scale at predetermined time intervals following treatment. The findings of this study may help clinicians select sealers based on their impact on postoperative pain and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with adequate oral hygiene.
* Teeth with no previous endodontic or restorative treatment.
* Teeth that do not respond to cold test and electric pulp test during vitality assessment.
* Teeth that are asymptomatic prior to treatment.
* Mandibular first or second molar teeth with complete root development.
* No bleeding observed in the pulp chamber after caries removal.
* Teeth with a Periapical Index (PAI) score of 3 or less.
* Patients who have not used antibiotics within the last 1 month.
* Patients who have not used analgesics within the last 72 hours.

Exclusion Criteria:

* Presence of systemic diseases that may affect healing (e.g., uncontrolled diabetes, immunosuppression).
* Pregnancy or breastfeeding.
* Teeth with a history of trauma, resorption, or previous endodontic access.
* Teeth with root canal calcifications or anatomical abnormalities preventing standard instrumentation.
* Presence of sinus tract, swelling, or acute apical abscess.
* Teeth with a Periapical Index (PAI) score greater than 3.
* Patients taking medications that may alter pain perception (e.g., corticosteroids, neuropathic pain medications).
* Patients unable to comply with follow-up pain recordings.
* Patients with known allergy to any materials used in the study (e.g., sodium hypochlorite, sealers).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Level | First 7 days after treatment (24 hours, 48 hours, 72 hours, and 7 days)
  Postoperative pain will be recorded using a 10-cm Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain. Participants will report their pain levels at 24 hours post-treatment, 48 hours post-treatment, 72 hours post-treatment, and on 7 days post-treatment following single-visit root canal treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Dentistry, Erzurum, palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No